CLINICAL TRIAL: NCT00052949
Title: Phase II Trial of STI571 in Patients With Relapsed Small Cell Lung Cancer
Brief Title: Imatinib Mesylate in Treating Patients With Recurrent Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01801; NCI-2012-01801 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000269156; NCCTG-N0124; CALGB-30201; N0124 (Other: North Central Cancer Treatment Group); N0124 (Other: CTEP); U10CA025224 (NIH)
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Recurrent Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Imatinib Mesylate

ARMS (1):
- Treatment (imatinib mesylate) (Experimental): Patients receive oral imatinib mesylate twice daily for 28 days. Courses continue in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of imatinib mesylate in treating patients who have recurrent small cell lung cancer. Imatinib mesylate may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate, time to progression, and overall survival of patients with recurrent small cell lung cancer treated with imatinib mesylate.

II. Correlate the presence of c-Kit mutations in tumor tissue with treatment response in patients treated with this drug.

III. Correlate individual patient variation in clinical (toxicity and/or activity), pharmacologic (pharmacokinetic/pharmacodynamic parameters), and/or biologic (correlative laboratory study results) responses to this drug with genetic differences in proteins involved in drug response (transport, metabolism, and/or mechanism of action).

OUTLINE: This is a multicenter study. Patients are stratified according to length of prior therapy (less than 3 months vs at least 3 months).

Patients receive oral imatinib mesylate twice daily for 28 days. Courses continue in the absence of disease progression or unacceptable toxicity.

*Patients are followed every 3 months until disease progression and then every 6 months for up to 3 years after registration.

NOTE: *Patients who develop CNS metastasis as the only site of disease progression receive therapeutic whole-brain radiotherapy and then resume study therapy.

PROJECTED ACCRUAL: A total of 41 patients for stratum I will be accrued within 21 months and 50 patients for stratum II will be accrued within 25 months for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed small cell lung cancer (SCLC)

  * No mixed histology
* Must have received only 1 prior treatment regimen (e.g., cyclophosphamide, doxorubicin, and vincristine alternating with etoposide and cisplatin allowed)
* c-Kit positive by immunohistochemistry (at least 1+)
* At least 1 unidimensionally measurable lesion

  * Longest diameter at least 20 mm
* No uncontrolled CNS metastasis

  * Treated CNS metastasis allowed
* Performance status - ECOG 0-2
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL
* Total bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Direct bilirubin no greater than ULN
* Creatinine no greater than 1.5 times ULN
* No unstable angina pectoris
* No uncontrolled congestive heart failure within the past 3 months unless ejection fraction is greater than 40%
* No myocardial infarction within the past 3 months
* No uncontrolled infection
* No other malignancy within the past 3 years except skin cancer or localized prostate cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study participation
* See Disease Characteristics
* More than 3 weeks since prior chemotherapy
* More than 2 weeks since prior radiotherapy
* No concurrent radiotherapy(including palliative therapy for bone pain)

  * Concurrent whole-brain radiotherapy for CNS progression allowed
* More than 3 weeks since prior major surgery
* No prior imatinib mesylate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2003-05; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The proportion of patients progression-free | 16 weeks
  Ninety-five percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Survival time | From registration to death due to any cause, assessed up to 3 years
  Estimated using the method of Kaplan-Meier.
Time to disease progression | From randomization to documentation of disease progression, assessed up to 3 years
  Estimated using the method of Kaplan-Meier.
Duration of response (complete response [CR] or partial response [PR]) | The date from which the patient's objective status if first noted to be either a CR or PR to the date progression is documented, assessed up to 3 years
Time to treatment failure | From the date of registration to the date at which the patient is removed from treatment due to progression, toxicity, refusal, or death, assessed up to 3 years
Toxicity defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment, per the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 2.0 | Up to 3 years
  The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Adjei, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States